CLINICAL TRIAL: NCT06826911
Title: The Effect of Health Literacy of Teachers and Parents on the Quality of Life of Primary School Students
Status: Not yet recruiting | Type: Observational
Sponsor: Duzce University (Other)
Responsible Party: Sponsor
Other Study IDs: Duzce-U-merve0005
Record Dates: First submitted 2025-02-10; First posted 2025-02-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Health Literacy; Life Quality
Keywords: Health literacy; Life quality; Primary school students

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Parents: This group consists of parents of students studying in primary school. The Personal Information Form and the Turkey Health Literacy Scale will be completed by the parents.
- Students: This group consists of students studying in primary school. The Generic Health-Related Quality of Life Scale for Children (Kid-KINDL)will be completed for the student.
- Teachers: This group consists of teachers in primary school. The Teacher Personal Information Form and the Turkey Health Literacy Scale will be completed by the teachers.

SUMMARY:
Health literacy (HL) is defined by the World Health Organization as "the achievement of a level of knowledge, personal skills, and confidence to take action to improve individual and community health by changing lifestyle and living conditions". Health literacy encompasses various skills that enhance individuals' quality of life, such as accessing accurate health information, adopting healthy lifestyle behaviours, utilizing healthcare services, and making informed health-related decisions. To raise the health literacy of a society, it is essential first to identify and enhance the health literacy of the family, the smallest unit of society. Moreover, it is well-established that parents serve as role models in fostering positive health behaviours and improving the quality of life of their children.

Aim: The aim of this study is to determine the impact of the health literacy of teachers and parents, who are thought to influence school-age children's perceptions of health and life, on the quality of life of primary school students.

DETAILED DESCRIPTION:
Health literacy (HL) is defined by the World Health Organization as "achieving a level of knowledge, personal skills, and confidence to take action to improve individual and community health by changing lifestyle and living conditions". Health literacy is considered a concept encompassing various skills that enhance individuals' quality of life, such as accessing accurate health information, adopting healthy lifestyle behaviours, utilizing healthcare services, and making informed health-related decisions. To improve society's health literacy, it is crucial first to identify and develop the health literacy of the family, the smallest unit of society. Adult family members are not only responsible for their health but also for fostering their children's health behaviours and meeting their health needs. Parents are known to serve as role models in encouraging positive health behaviours and enhancing their children's quality of life. Low health literacy in adults is associated with adverse health outcomes. Parents who struggle to take responsibility for their health are likely to face challenges in addressing their children's health needs, which may lead to frequent health problems in children. Studies reveal that parents with low health literacy are insufficient in meeting their children's health needs, utilizing healthcare services, taking precautions against health risks, ensuring proper medication use and monitoring side effects, managing chronic illnesses, and encouraging their children to adopt healthy lifestyle behaviours. The school-age period is particularly significant as it is a critical phase of rapid social, physical, and cognitive development, shaping a healthy and successful society. Schools are central to children's social interactions, where they spend most of their time, and thus teachers play an important role as role models in their lives. Studies in our country indicate that teachers' health literacy levels are often insufficient.

The purpose of this study is to determine the impact of teachers' and parents' health literacy, thought to influence school-age children's perceptions of health and life, on the quality of life of primary school students. The study is expected to contribute to protecting public health, developing health services and policies aimed at improving the health literacy of parents and teachers and preventing health inequalities by enhancing students' quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Students, parents and teachers located at Uzun Mustafa Primary School in the city centre of Düzce.

  * Voluntary participation in the study.

Exclusion Criteria:

* Parents who do not agree to participate in the study and their children will be excluded from the research.
* Teachers who do not agree to participate.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study will be conducted at Uzun Mustafa Primary School, affiliated with the Ministry of National Education, in the city centre of Düzce between December 2024 and June 2025. A total of 52 teachers working at Uzun Mustafa Primary School, along with 1,151 students and their parents, will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 2355 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Health literacy | one day
  The Turkey Health Literacy Scale was developed by Okyay and Abacıgil in 2016 to assess health literacy, in line with the European Health Literacy Research Consortium. The scale consists of 32 questions. It has a 2x4 matrix structure, with two dimensions (treatment and services, and disease prevention/health promotion) and four processes (accessing health-related information, understanding health-related information, evaluating health-related information, and using/applying health-related information), making a total of eight components. The Cronbach's Alpha value of the scale is 0.927. The scale is rated as follows: "1. Very Easy, 2. Easy, 3. Neither easy nor difficult, 4. Difficult, 5. Very Difficult." The health literacy level is categorized into four groups based on the score obtained: (0-25) points: Inadequate health literacy, (>25-33) points: Problematic - limited health literacy, (>33-42) points: Adequate health literacy, (>42-50) points: Excellent health literacy.
The Generic Health-Related Quality of Life Scale for Children | one day
  The Kid-KINDL (8-12 years) is a general-purpose (generic) quality-of-life scale designed for children. It consists of 24 items and 6 dimensions: physical well-being, emotional well-being, self-esteem, family, friends, and school. Originally developed in German, the KINDL has been translated into 14 languages. Each dimension comprises 4 items. While scores for each dimension are calculated independently, a total health-related quality of life (HRQoL) score is also derived from the combination of these six dimensions. The Kid-KINDL items are rated using a 5-point Likert scale ranging from 1 (never) to 5 (always). Negative items (questions 1, 2, 3, 6, 7, 8, 15, 16, 20, and 24) are reverse-coded for scoring. To calculate scores: Responses for each dimension are summed. The scores are transformed to a 0-100 scale for standardization. A higher score indicates a better quality of life. This scale is widely used to evaluate children's perspectives on their health and overall quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Merve Cakar, PhD, Principal Investigator — Duzce University
Locations (1):
- Duzce University, Düzce, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No